CLINICAL TRIAL: NCT04545112
Title: Prospective, Non-randomized, First in Human (FIH) Clinical Study to Assess the Feasibility of the Novel Xeltis Coronary Artery Bypass Graft (XABG)
Brief Title: Xeltis Coronary Artery Bypass Graft (XABG) First in Human (FIH)
Acronym: XABG FIH
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Xeltis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XEL-CR-07
Record Dates: First submitted 2020-08-28; First posted 2020-09-10 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-02

CONDITIONS: Multi Vessel Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- XABG (Experimental)
  Interventions: Device: CABG

INTERVENTIONS:
Device: CABG — Elective, coronary artery bypass (CABG) surgery. Each study subject will receive an left internal mammary artery (LIMA) conduit to the left anterior descending (LAD) coronary artery. Patients with uncompromised saphenous veins will receive a SVG to the LCX or RCA and the XABG to the remaining territory. Patients with compromised arterial and/or saphenous veins, (i.e., "no-vein" patients), will receive one XABG to the LCX or RCA to achieve incomplete revascularization.

SUMMARY:
A prospective, single arm, non-randomized FIH feasibility study to evaluate the preliminary safety and performance of the XABG technology in patients with multi-vessel atherosclerotic coronary artery disease, scheduled by the local Heart Team to undergo elective coronary artery bypass (CABG) surgery.

ELIGIBILITY:
Inclusion Criteria:

* All gender, 18 years of age or older with a minimum life expectancy of 2 years.
* Elective multi-vessel atherosclerotic CAD patients, selected and accepted by the local Heart Team and confirmed by the Screening Committee for CABG surgery.
* LIMA bypass graft to LAD coronary artery indicated and feasible.
* XABG target vessel(s) with proximal occlusion and/or critical stenosis. and with a diameter of ≥ 2 mm and sufficient distal run-off (thrombolysis in myocardial infarction risk (TIMI)-Score ≥ 2).
* Patient has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent.
* Patient has been informed and agrees to pre- and post-procedure follow-up, including follow-up CT scan and coronary angiogram.
* Patient is suitable for percutaneous coronary intervention (PCI) procedures in case of required emergent procedures at discretion of the local Heart Team.

Exclusion Criteria:

* Total arterial bypass grafting indicated and feasible
* Any previous open-heart surgery or surgical/transcatheter procedure that could compromise imaging follow up.
* History of cardiac resynchronization therapy (CRT) or implantable cardioverter defibrillator (ICD) implantation
* Concomitant cardiac surgery (e.g. valve treatment, ablation).
* Myocardial infarction (MI) within 21 days or cerebral vascular accident (CVA) within 90 days prior to the CABG procedure
* Left ventricular ejection fraction ≤ 35%.
* Severe kidney disease, renal dysfunction (Cr> 2.0mg/dL) or Glomerular Filtration Rate (GFR) < 50mL/min or active dialysis patients.
* Moderate to severe chronic obstructive pulmonary disease (COPD) with a forced expiratory volume (FEV) <1.5 lit/sec.
* Endocarditis, pericarditis or any other active systemic infection that would interfere with subject safety.
* Active bleeding disorder and/or any coagulopathy or thromboembolic disease or other indication requiring anticoagulation
* Known Heparin Induced Thrombocytopenia (HIT)
* Abnormal blood values (e.g. leukopenia, anemia or thrombocytopenia) that could influence graft hemostasis or patient recovery.
* Use of immunosuppressive therapy or medication or active clinically inflammatory/autoimmune disease or immunodeficiency that likely interferes with restorative therapies
* Known and non-treatable allergies to study device (Nitinol) or agents/medication, such as contrast agents, antiplatelet therapy, beta-blocker, statins required for study assessment or optimal post-CABG medical treatment (hospital SOC).
* Need for emergency surgery for any reason and/or intervention/surgery prior to and within 12 months after the CABG surgery that requires antiplatelet therapy discontinuation.
* Currently in investigational device or drug study or participated in the last 30 days.
* Pregnancy or females currently lactating or childbearing potential who are sexually active and are not willing to use adequate contraceptive precautions for the next 2 years.
* Subject has medical, social or psychosocial factors that, in the opinion of the Investigator, could impact safety or compliance.
* Has any other condition, in the opinion of the principal investigator, which would put the patient at increased risk from participating in the study or otherwise prevent participation.

Intra-operative Exclusion Criteria:

* Severe calcified aorta (porcelain aorta) or diseased aorta that precludes proximal vein graft anastomoses
* Unsuccessful LIMA to LAD anastomosis
* After chest opening and visual inspection identification of active pericarditis/endocarditis and/or diffuse calcification in target vessels and/or any other reason precluding sufficient distal anastomoses.
* Smaller distal coronary artery and/or poor distal run-off and/or XABG patient/device size mismatch as initially expected in the pre-operative workup.
* Hemodynamic instability before XABG attempt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2031-02-15 (Estimated)

PRIMARY OUTCOMES:
Procedural success during the first 30 days | 30 days
  XABG technology performs as intended with successful proximal and distal anastomoses and graft patency at the conclusion of the procedure and at 30 days. Patency is defined as a diameter stenosis less than 50%
Freedom from device related Serious Adverse Events (SAEs) | 30 days

SECONDARY OUTCOMES:
Intimal hyperplasia area | 12 months
  Assessed by OCT
Graft patency | 30 days, 6 months, 12 months
  Patency defined as a diameter stenosis less than 50%
Lumen diameter uniformity | 30 days, 6 months, 12 months
  Using Fitzgibbon's 3-point ordinal uniformity scale
Freedom from Major Adverse Cardiac and Cerebrovascular Events (MACCE) | 30 days, 6 months, 12 months, and yearly until 5 years
  Absence of device related SAEs
Freedom from vein harvesting related wound infection, non-infective wound healing disturbances, and leg pain | 30 days and 6 months
  Leg pain will be assessed by standard 10-point VAS scale and presented as descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Bart Meuris, MD, Principal Investigator — UZ Leuven
Locations (4):
- UZ Leuven, Leuven, Belgium
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- Poland (2):
  - John Paul II Hospital Krakow, Krąków
  - Medicover Hospital, Warsaw